CLINICAL TRIAL: NCT00463697
Title: A Randomized, Single-dose, Dose-ascending, Double Blind, Placebo-controlled, 5-way Crossover Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Inhaled Doses of GW642444M With Magnesium Stearate in Asthmatic Patients
Brief Title: A Study To Investigate The Effect Of Inhaling A Single Dose Of GW642444M In Asthmatic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2C106996
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GW642444,; magnesium stearate,; asthmatic patients
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- GW642444M 25mcg (Experimental): Subject will inhale single dose of GW642444M 25 mcg via a DISKUS device in morning.
  Interventions: Drug: GW642444M (25, 100 & 400 mcg)
- GW642444M 100mcg (Experimental): Subject will inhale single dose of GW642444M 100 mcg via a DISKUS device in morning.
  Interventions: Drug: GW642444M (25, 100 & 400 mcg)
- GW642444M 400mcg (Experimental): Subject will inhale single dose of GW642444M 400 mcg via a DISKUS device in morning.
  Interventions: Drug: GW642444M (25, 100 & 400 mcg)
- GW642444H 100mcg (Experimental): Subject will inhale single dose of GW642444H 100 mcg via a DISKUS device in morning.
  Interventions: Drug: GW642444H (100mcg)
- placebo (Placebo Comparator): Subject will inhale single dose of Placebo via a DISKUS device in morning.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GW642444H (100mcg) — H salt
  Arms: GW642444H 100mcg
Drug: placebo — placebo
  Arms: placebo
Drug: GW642444M (25, 100 & 400 mcg) — M salt
  Other Names: placebo; GW642444M (25; 100 & 400 mcg); GW642444H (100mcg)
  Arms: GW642444M 100mcg; GW642444M 25mcg; GW642444M 400mcg

SUMMARY:
This study will involve the use of a new compound, GW642444 that is being developed for the treatment of asthma and chronic obstructive pulmonary disease (COPD). It works by acting on cells in the lungs, causing some of the muscles around the lungs to relax and open up better (bronchodilation), making breathing easier. When a medicine is made into a form ready to be given to patients, the active ingredient is often prepared with another ingredient called a salt to help make it stable, and inactive ingredients are often added. Inactive ingredients might be used to help a medicine work better, to make it easier to produce the medicine, or to make it easier to get an accurate dose of medicine. In previous studies the study drug has been given as a dry powder containing either the "H" salt (with the inactive ingredient lactose), or containing the "M" salt (with the inactive ingredients lactose and cellobiose octaacetate). The "M" salt form of the study drug has been altered to contain lactose and a new inactive ingredient called magnesium stearate (instead of cellobiose octaacetate).

Participants in this study will receive both the "H" salt (GW642444H) and the new "M" salt (GW642444M) containing magnesium stearate. This study will be the first time the new "M" salt form of the study drug will be given to asthmatic patients.

ELIGIBILITY:
Inclusion criteria:

* male or female (of non-childbearing potential) between 18 - 70 years
* History of stable mild to moderate asthma
* non - smokers
* currently taking daily doses of inhaled fluticasone propionate 200 - 500 mcg (or equivalent)
* body weight >50 kg with BMI 19-29.9 kg/m2
* normal ECG assessment

Exclusion criteria:

* history of significant disease
* history of life threatening asthma
* recent respiratory tract infection
* recent change of asthma medication
* treatment with high dose inhaled corticosteroids or oral corticosteroids
* recent participation in another trial
* history of drug or alcohol abuse
* known allergies (excluding asthma)
* recent blood donation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-04-02 (Actual); Primary Completion 2007-08-04 (Actual); Study Completion 2007-08-04 (Actual)

PRIMARY OUTCOMES:
General safety and tolerability of the new formulation of GW642444 as measured by ECG, blood pressure, pulse rate and blood and urine tests. Serial measurements are made over 24 hours on 5 separate occasions (separated by 1 - 2 weeks). | Serial measurements are made over 24 hours on 5 separate occasions (separated by 1 - 2 weeks).

SECONDARY OUTCOMES:
Airways relaxation assessed by lung function tests. Effect of study medicine on the body and amount of medicine in the body measured by potassium, glucose and medicine in blood samples. Measurements made over 24 hours on 5 occasions (1-2 weeks apart). | Measurements made over 24 hours on 5 occasions (1-2 weeks apart).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United Kingdom (3):
  - GSK Investigational Site, Harrow, Middlesex
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kempsford R, Norris V, Siederer S. Vilanterol trifenatate, a novel inhaled long-acting beta2 adrenoceptor agonist, is well tolerated in healthy subjects and demonstrates prolonged bronchodilation in subjects with asthma and COPD. Pulm Pharmacol Ther. 2013 Apr;26(2):256-64. doi: 10.1016/j.pupt.2012.12.001. Epub 2012 Dec 8. PMID 23232038
- See also: Results for study B2C106996 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/B2C106996?search=study&search_terms=B2C106996#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: B2C106996 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: B2C106996 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: B2C106996 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: B2C106996 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: B2C106996 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: B2C106996 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: B2C106996 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register